CLINICAL TRIAL: NCT00951249
Title: Feasibility Study of a Community-Level, Multi-Component Intervention for Black Men Who Have Sex With Men
Brief Title: Feasibility Study of a Multi-Component Intervention for Black Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 061; 1U01AI068619 (NIH)
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: HIV Infections
Keywords: MSM; HIV infections; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Mass Screening; Counseling

ARMS (1):
- A (Experimental): HIV-infected and uninfected black MSM
  Interventions: Behavioral: Referral of Partners; Behavioral: Screening for STIs and counseling; Behavioral: Peer health care system navigators; Behavioral: Enhanced counseling

INTERVENTIONS:
Behavioral: Referral of Partners — Referral of up to five sexual partners by index participants for enrollment into the study
Behavioral: Screening for STIs and counseling — Identification of STIs and treatment or referral for treatment, if applicable
Behavioral: Peer health care system navigators — HIV/STI treatment and other medical and social services
Behavioral: Enhanced counseling — Counseling and referral for care offered to participants for issues such as substance use and mental health

SUMMARY:
It has been estimated that black men who have sex with men (MSM) account for one quarter of all new HIV infections in the US annually, yet little prevention work has been directed towards this population. The purpose of this study is to research and potentially design a new and better way to try and slow the spread of HIV among black MSM.

DETAILED DESCRIPTION:
In the US, men who have sex with men (MSM) comprise the largest proportion of new HIV infections, with black MSM being infected at significantly higher rates. Differences in sexual-risk behaviors and substance use do not explain the disproportionate HIV rates by race among MSM. The most likely explanations are low frequency of HIV testing, high HIV prevalence within sexual networks, high prevalence of other sexual transmitted infections (STIs), and barriers to health care access and HIV/STI treatment. These result in later diagnoses of HIV-infected men, more frequent STIs, and fewer HIV-infected men having access to care.

The purpose of this study is to gather information on the achievability and acceptability of the following interventions:

A.) Referral of up to five sexual partners by index participants for enrollment into the study B.) Counseling and testing for HIV C.) Counseling and testing for other STIs D.) Counseling and referral for care offered to participants for issues such as substance use and mental health.

E.) Engagement with peer health care system navigators (PHNs) to facilitate uptake of health care and other services.

These interventions are designed to impact several factors related to the HIV epidemic among black MSM. At the individual level, the interventions will address personal risk factors for either acquiring or transmitting HIV, including identifying undiagnosed HIV or STI infections, and helping participants to reduce risk-behaviors, such as those influenced by drugs and alcohol. The interventions are also designed to have an impact at the population level. If successful, they will lower the viral load in HIV-infected men by identifying those who qualify for HIV treatment and intervening to increase treatment and access to healthcare. Overall, the study investigators propose that by lowering both the proportion of men with undiagnosed HIV infection and those with chronic, untreated infection, the rates of HIV transmission will be reduced among the black MSM population. This is a feasibility study, designed to provide estimates about the potential effectiveness of these interventions. These estimates will then be used to determine whether a large-scale trial of the interventions would be successful.

Approximately 2418 total participants will be enrolled into the study at six different sites. Participants will be enrolled in one of two ways: either directly from the community, or referred by other participants (sexual network partners). The total duration of the study will be two years. This includes 12 months for participant accrual and 12 months of follow-up for each participant. All participants will have an enrollment visit, during which he will complete a questionnaire covering topics such as sexual risk behaviors, drug and/or alcohol use, current and prior engagement with the health care system, barriers to HIV care, unmet service needs, frequented venues, attitudes about race, sexual history, research, and health care. Participants will also be asked to enumerate 5 social and 10 sexual network members (age, race, HIV status), information which will be used to better understand the characteristics of black MSM social and sexual networks.

Participants will be offered HIV and STI testing and counseling. Those with reactive HIV rapid test results will have HIV infection confirmed by Western blot and will have a CD4 cell count and viral load test performed. Counselors will provide post-test HIV participants counseling to those who have had HIV rapid test performed and will schedule all participants to return to the clinic approximately two weeks later to receive additional test results. The counselor will also discuss the participant's engagement in health care, and will determine the participant's health and other service needs. The counselor will also inquire about homophobic or partner violence and provide any care referrals if needed. Additionally, risk reduction counseling will be provided.

Study participation will end after the initial visit for three groups of participants. These groups include those who have: A.) an HIV-positive diagnosis prior to screening for this study and are either in care (have seen a health care provider for HIV-related care in the last six months)or who have unprotected sex only with HIV-infected partners. B.) HIV-uninfected participants enrolled after the site's 200 person cap for this category, and C.) participants who refuse HIV testing after the site's fist 20 participants in this category have been enrolled. Participants who fall into the categories listed above will provide only baseline cross-sectional data.

All other participants will then have the counselor explain about peer health care system navigation and introduce the participant to the PHN. The PHN will meet with the participant and schedule an initial discussion, unless the participant does not have any need for the navigation, in which case the PHN will plan to call after a few weeks to check for any emerging needs. The PHN will interact with the participant on a schedule that is independent of the study visit schedule and is determined by the participant's needs. The PHN's role will be to help the participant overcome his barriers to health care through a number of activities.

Follow-up visits are scheduled infrequently, so participants may be contacted periodically between visits to stay in touch and provide updated locator information. Visits will include the completion of a questionnaire, HIV testing for those who were not infected at the prior visit, with confirmation and follow-up tests if necessary. A viral load test will be performed for HIV-infected participants at the time of diagnosis and again at 52 weeks. All participants will receive STI counseling and testing at 26 and 52 weeks. Participants will receive counseling to include risk reduction counseling and pre- and post- test counseling, as needed. Participants will also be counseled for issues such as mental health and substance use and referred for care as appropriate. Participants will be asked to report any STI or HIV diagnoses they receive between visits and to provide documentation of diagnoses. Plasma specimens for testing will also be collected from all participants at all visits.

In order to collect additional information on the black MSM population, interviews and focus groups will also be a component in this study. Focus group meetings will be approximately 1.5 to 2 hours long and will be conducted at locations that allow for privacy and confidentiality. Interviews will last for between 60 to 90 minutes and will be conducted with individual participants. Interviews will be audio recorded and transcribed.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Black, African American, Caribbean Black, or multiethnic Black
* At least one instance of unprotected anal intercourse (UAI) with a man in the past six months
* Residing in the metropolitan area and do not plan to move away during the time of study participation

Exclusion Criteria:

* Co-enrollment in any other HIV interventional research study or have been enrolled in an HIV vaccine trial in which they were either in the active arm or do not know the arm in which they were enrolled.
* Would be enrolled as a community-recruited participant in a category that has already reached its enrollment cap
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1553 (Actual)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of participants enrolled at each city | At 52 Weeks
Proportion of participants who agree to HIV testing | Throughout study
Proportion of participants who agree to STI testing | Throughout study
Proportion of participants who use PHN | Throughout study
Proportion of participants who are newly diagnosed with HIV at enrollment | At Study Entry
Increase in condom use | Study Entry to Week 52
Decrease in viral load among HIV-infected participants who initiate HAART during their study participation | At Week 52
Decrease in STI | At Study Entry to Week 52

SECONDARY OUTCOMES:
Number of participants with recent HIV infection | At Study Entry
Number of participants with acute HIV infection | At Week 52
Number of seroconversions during follow-up among those who are HIV-uninfected | At Follow-up
Number of sex partners | At Study Entry, and Weeks 26 and 52
Number of sero-discordant or sero-unknown partners | At Study Entry, and Weeks 26 and 52
Type and frequency of anal intercourse | At Study Entry, and Weeks 26 and 52
Level of condom use | At Study Entry, and Weeks 26 and 52
Partner change rate | At Study Entry, and Weeks 26 and 52
As individually self-reported by participants: network size, composition, density, multiplexity, durability, and homogeneity | Throughout study
Overlap of participant's sexual network with his social network | Throughout study
Attitudes of black MSM toward other prevention interventions | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Beryl Koblin, PhD, Study Chair — New York Blood Center; Kenneth Mayer, MD, Study Chair — Fenway Community Health Center; Darrell P. Wheeler, PhD, MPH, ACSW, Study Chair — School of Social Work, Hunter College
Locations (8):
- United States (8):
  - UCLA Vine Street CRS, Los Angeles, California
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - George Washington University, Washington D.C., District of Columbia
  - The Ponce de Leon Ctr. CRS, Atlanta, Georgia
  - Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - The Fenway Institute, Boston, Massachusetts
  - NY Blood Ctr./Union Square CRS, New York, New York
  - Harlem Hospital Center/Columbia University CRS, New York, New York

REFERENCES:
- [Background] Bissessor M, Fairley CK, De Guingand D, Bradshaw CS, Chen MY. Delay in the diagnosis of early syphilis among men who have sex with men: need for greater community and health provider education. Int J STD AIDS. 2009 Jan;20(1):52-3. doi: 10.1258/ijsa.2008.008254. PMID 19103894
- [Background] Rowniak S. Safe sex fatigue, treatment optimism, and serosorting: new challenges to HIV prevention among men who have sex with men. J Assoc Nurses AIDS Care. 2009 Jan-Feb;20(1):31-8. doi: 10.1016/j.jana.2008.09.006. PMID 19118769